CLINICAL TRIAL: NCT05435313
Title: A Single-center, Single-arm, Open-label Clinical Study of Fruquintinib Combined With Tislelizumab and HAIC in Patients With Advanced Colorectal Liver Metastases Cancer Who Failed Standard Therapy
Brief Title: Fruquintinib Combined With Tislelizumab and HAIC in Patients With Advanced Colorectal Liver Metastases Cancer Who Failed Standard Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C122
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; tislelizumab; raltitrexed; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy (Experimental): Combination: Fruquintinib plus Tislelizumab and HAIC (TOMOX/TOMIRI)
  Maintenance: Fruquintinib plus Tislelizumab
  Interventions: Procedure: HAIC; Drug: Fruquintinib; Drug: Tislelizumab; Drug: Raltitrexed; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Procedure: HAIC — After successful percutaneous hepatic artery cannulation, superior mesenteric arteriogram and hepatic arteriogram were performed, and after confirming that the subjects were eligible for enrollment according to the results, the hepatic artery was cannulated to the predetermined position. The catheter was connected to a syringe pump in the ward for continuous pumping of drugs.
Drug: Fruquintinib — 3mg, qd, po, 21 days for a cycle, Suspend medication on the day of HAIC
Drug: Tislelizumab — 200mg, ivgtt, d1, 21 days for a cycle
Drug: Raltitrexed — 2 mg/m2, hepatic artery infusion for 15 min, d1, 4-6 Cycles
Drug: Oxaliplatin — 85 mg/m2, hepatic artery infusion for 2 h, d1, 4-6 Cycles
Drug: Irinotecan — 120mg/m2, hepatic artery perfusion for 30-90min, d1, 4-6 Cycles

SUMMARY:
This is a single-center, single-arm, open-label clinical study, to explore the efficacy and safety of fruquintinib combined with tislelizumab and HAIC (hepatic arterial infusion chemotherapy) in patients with colorectal liver metastases cancer (CRLM) who failed standard therapy.

DETAILED DESCRIPTION:
Liver is the most common metastatic site in patients with colorectal cancer (CRC) and the leading cause of death in patients. Surgery is the best way to cure CRLM, but few patients can receive surgery, and patients prone to recurrence after surgery. It is an urgent topic to choose an effective treatment method with less side effects for CRLM patients. HAIC is a unique and effective treatment option for CRLM patients. Fruquintinib is a small molecule angiogenesis inhibitor, and has been recommended for third-line treatment of metastatic colorectal cancer (mCRC). Tislelizumab is a humanized IgG4 anti-PD-1 monoclonal antibody, meanwhile, tislelizumab shows significant and durable antitumor activity in patients with CRC, and is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed
2. Histologically or cytologically confirmed unresectable advanced colorectal liver metastases cancer
3. Age ≥ 18 years, ≤75 years
4. ECOG PS：0-1
5. Expected overall survival ≥3 months
6. Patients must have at least one measurable liver metastases (RECIST 1.1)
7. Patients who have previously failed standard treatment, or who cannot tolerate standard treatment
8. Patients must have adequate organ and bone marrow function
9. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration

Exclusion Criteria:

1. Patients who are allergic or suspected to be allergic to the study drug or similar drugs
2. Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
3. Participating in other clinical trials and received at least one treatment within 4 weeks before enrollment
4. Patients with autoimmune disease or history of autoimmune disease within 4 weeks before enrollment
5. patients currently have central nervous system (CNS) metastasis or previous brain metastasis and the symptom control time is less than 2 months
6. Patients cannot take fruquintinib orally
7. Patients who have received organ transplantation and bone marrow transplantation in the past
8. Have taken other strong inducers or inhibitors of CYP3A4, P-gp substrates and BCRP substrates within 2 weeks before the First medication
9. Received any operation (except biopsy) or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before enrollment
10. Pleural effusion or ascites causing relevant clinical symptoms, including respiratory syndrome (dyspnea≥CTC AE grade 2)
11. Clinically significant electrolyte abnormality；
12. Systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs; Or patients need more than two antihypertensive drugs
13. Proteinuria ≥ 2+ (1.0g/24hr);
14. Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI, or other conditions that may cause GI bleeding and perforation as determined by the investigator;
15. Have evidence or history of bleeding tendency within 3 months or thromboembolic events within 12 months before enrollment
16. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; NYHA classification > 2 Grade; ventricular arrhythmia requiring medical therapy; ECG showing QTc interval ≥ 480 ms
17. Active or uncontrolled serious infection (≥CTCAE grade 2 infection)
18. Pregnant or lactating women
19. Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the judgment of investigator that the patient is not suitable for the the study drug (such as having epileptic seizures and require treatment), or would affect the interpretation of study results, or put patients at high risk
20. Clinical uncontrolled active infections, including human immunodeficiency virus (HIV) infection, active hepatitis B / C (HBV DNA Positive[1×104 copies/mL or >2000 IU/ml], HCV RNA positive[>1×103 copies/mL]);
21. Patients have other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental diseases) that require concomitant treatment, and serious laboratory abnormalities. Accompanied by family or social factors, which will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Progression-Free Survival rate at 6 months | 6 months
  The proportion of patients who did not experience disease progression or death from treatment initiation to 6 months
overall survival (OS) | 24 months
  OS is the time from enrollment to death due to any cause.
Adverse events as assessed by NCI CTCAE v5.0 | 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China